CLINICAL TRIAL: NCT01557504
Title: A Study to Assess the Pharmacokinetics and the Ability for Pediatric Patients With Type 2 Diabetes to Swallow MK-0431A XR Tablets
Brief Title: A Study to Assess the Pharmacokinetics and the Ability for Pediatric Participants With Type 2 Diabetes to Swallow MK-0431A XR Tablets (MK-0431A-296)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431A-296; 2020-003731-22 (EudraCT Number); MK-0431A-296 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Metformin; Thyroid Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin/metformin XR followed by placebo (Experimental): Day 1 (Period 1): participants will receive a single dose of two sitagliptin/metformin XR tablets with a low- to moderate-fat meal (breakfast). Days 2-4 (Period 1): participants will receive a single dose of two matching placebo tablets. Days 5-9 (Period 2): participants will receive a single dose of two matching placebo tablets with the evening meal.
  Interventions: Drug: Sitagliptin/metformin XR; Drug: Placebo; Drug: Metformin; Drug: Thyroid hormone
- Placebo only (Placebo Comparator): Days 1-4 (Period 1): participants will receive a single dose of two matching placebo tablets. Days 5-9 (Period 2): participants will receive a single dose of two matching placebo tablets with the evening meal.
  Interventions: Drug: Placebo; Drug: Metformin; Drug: Thyroid hormone

INTERVENTIONS:
Drug: Sitagliptin/metformin XR — Fixed dose combination tablet of immediate-release sitagliptin 50 mg and extended-release (XR) metformin 1000 mg (total daily dose, sitagliptin 100 mg and metformin XR 2000 mg).
  Other Names: MK-0431A XR; Janumet XR
  Arms: Sitagliptin/metformin XR followed by placebo
Drug: Placebo — Matching placebo to fixed dose combination tablet of sitagliptin and metformin. Matching placebo tablets are same size, shape and color as the active product, but do not contain any markings.
Drug: Metformin — Concomitant use of metformin is permitted during the study provided the participant has been receiving a stable metformin dose for at least 12 weeks prior to the dose of study drug. Administration of metformin will be withheld for 24 hours prior to study drug administration and for 24 hours postdose.
Drug: Thyroid hormone — Concomitant use of thyroid hormone (eg, levothyroxine) is permitted during the study provided the participant has been receiving a stable dose for at least 12 weeks prior to study drug administration and is euthyroid as documented by thyroid stimulating hormone testing at prestudy. Administration of thyroid hormone will be withheld for 24 hours prior to study drug administration and for 24 hours postdose.

SUMMARY:
The purpose of this study is to assess:

1. the safety and tolerability of two sitagliptin 50 mg/metformin 1000 mg XR tablets in pediatric participants with type 2 diabetes mellitus (T2DM), aged 10 to 17 years
2. the ability of pediatric participants with T2DM, aged 10 to 17 years, to swallow two sitagliptin 50 mg/metformin 1000 mg XR tablets or two matching placebo tablets (excluding marking)
3. the pharmacokinetics of sitagliptin and metformin following the administration of two sitagliptin 50 mg/metformin 1000 mg XR tablets to pediatric participants with T2DM, aged 10 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Female participant of reproductive potential must not be pregnant and agrees to use (and/or have their partner use) two acceptable methods of birth control
* T2DM diagnosed by American Diabetes Association criteria
* No clinically significant abnormality on electrocardiogram
* No clinical or laboratory evidence to indicate a diagnosis of type 1 diabetes
* Nonsmoker

Exclusion Criteria:

* Mental or legal incapacitation
* Estimated creatinine clearance of 80 mL/min or lower
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic disease
* Unable to refrain from or anticipates the use of any medication (with the exception of metformin and thyroid hormone) from approximately 2 weeks before the first dose of study drug through the poststudy visit
* Consumes alcohol or consumes excessive amounts of coffee, tea, cola, or other caffeinated beverages
* Had surgery, donated or lost 1 unit of blood, or participated in another investigational study within the past 4 weeks
* History of multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Currently a regular user (including illicit drugs) or has a history of drug (including alcohol) abuse
* Lactose intolerant

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2012-07-18 (Actual); Primary Completion 2014-04-29 (Actual); Study Completion 2014-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431A-296&kw=0431A-296&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin/Metformin XR Followed by Placebo: Day 1 (Period 1): participants received a single dose of two sitagliptin/metformin XR tablets with a low- to moderate-fat meal (breakfast). Days 2-4 (Period 1): participants received a single dose of two matching placebo tablets. Days 5-9 (Period 2): participants received a single dose of two matching placebo tablets with the evening meal.
- Placebo: Days 1-4 (Period 1): participants received a single dose of two matching placebo tablets. Days 5-9 (Period 2): participants received a single dose of two matching placebo tablets with the evening meal.
Period: Overall Study
Arm/Group | Sitagliptin/Metformin XR Followed by Placebo | Placebo
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Metformin XR Followed by Placebo | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Customized [Count of Participants; unit: Participants]
  10-13 years | 4 | 3 | 7
  14-17 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Successfully Swallowed Study Medication (Med) on Day 2
Description: The Swallowing Ability Questionnaire was completed on Day 2 after the participant received two matching placebo tablets (excluding marking) following consumption of a low- to moderate-fat meal in pediatric participants aged 10 to 17 years. The questionnaire consisted of five parts: could only swallow study med with help, easy to start swallowing study med, easy to swallow study med, felt like study med got stuck in throat, and had to swallow study med more than once. The number of participants who strongly agreed or agreed in each of the five parts is reported.
Time Frame: Day 2
Population: Per protocol population defined as all participants who completed at least one period of treatment and had available data. On Day 2, all participants received matching placebo, so the two treatment groups were pooled on Day 2.
Measure: Number; unit: Participants
Groups:
- All Treated Participants: All participants who completed at least one period of treatment and had available data. All participants received a single dose of two matching placebo tablets on Day 2.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 24
Participants
  Strongly Agreed: Could Only Swallow Med With Help | 6
  Agreed: Could Only Swallow Med With Help | 7
  Strongly Agreed: Easy to Start Swallowing Med | 10
  Agreed: Easy to Start Swallowing Med | 12
  Strongly Agreed: Easy to Swallow Med | 13
  Agreed: Easy to Swallow Med | 10
  Strongly Agreed: Felt Like Med Got Stuck in Throat | 0
  Agreed: Felt Like Med Got Stuck in Throat | 4
  Strongly Agreed: Had to Swallow Med More Than Once | 2
  Agreed: Had to Swallow Med More Than Once | 3

2. Primary Outcome: Number of Participants Who Successfully Swallowed Study Med on Day 4
Description: The Swallowing Ability Questionnaire was completed on Day 4 after the participant received two matching placebo tablets (excluding marking) following consumption of a low- to moderate-fat meal in pediatric participants aged 10 to 17 years. The questionnaire consisted of five parts: could only swallow study med with help, easy to start swallowing study med, easy to swallow study med, felt like study med got stuck in throat, and had to swallow study med more than once. The number of participants who strongly agreed or agreed in each of the five parts is reported.
Time Frame: Day 4
Population: Per protocol population defined as all participants who completed at least one period of treatment and had available data. On Day 4, all participants received matching placebo, so the two treatment groups were pooled on Day 4.
Measure: Number; unit: Participants
Groups:
- All Treated Participants: All participants who completed at least one period of treatment and had available data. All participants received a single dose of two matching placebo tablets on Day 4.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 24
Participants
  Strongly Agreed: Could Only Swallow Med With Help | 6
  Agreed: Could Only Swallow Med With Help | 6
  Strongly Agreed: Easy to Start Swallowing Med | 8
  Agreed: Easy to Start Swallowing Med | 14
  Strongly Agreed: Easy to Swallow Med | 8
  Agreed: Easy to Swallow Med | 15
  Strongly Agreed: Felt Like Med Got Stuck in Throat | 0
  Agreed: Felt Like Med Got Stuck in Throat | 4
  Strongly Agreed: Had to Swallow Med More Than Once | 0
  Agreed: Had to Swallow Med More Than Once | 5

3. Primary Outcome: Number of Participants Who Successfully Swallowed Study Med on Day 6
Description: The Swallowing Ability Questionnaire was completed on Day 6 after the participant received two matching placebo tablets (excluding marking) following consumption of a low- to moderate-fat meal in pediatric participants aged 10 to 17 years. The questionnaire consisted of five parts: could only swallow study med with help, easy to start swallowing study med, easy to swallow study med, felt like study med got stuck in throat, and had to swallow study med more than once. The number of participants who strongly agreed or agreed in each of the five parts is reported.
Time Frame: Day 6
Population: Per protocol population defined as all participants who completed at least one period of treatment and had available data. On Day 6, all participants received matching placebo, so the two treatment groups were pooled on Day 6.
Measure: Number; unit: Participants
Groups:
- All Treated Participants: All participants who completed at least one period of treatment and had available data. All participants received a single dose of two matching placebo tablets on Day 6.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 24
Participants
  Strongly Agreed: Could Only Swallow Med With Help | 5
  Agreed: Could Only Swallow Med With Help | 7
  Strongly Agreed: Easy to Start Swallowing Med | 10
  Agreed: Easy to Start Swallowing Med | 11
  Strongly Agreed: Easy to Swallow Med | 11
  Agreed: Easy to Swallow Med | 12
  Strongly Agreed: Felt Like Med Got Stuck in Throat | 0
  Agreed: Felt Like Med Got Stuck in Throat | 3
  Strongly Agreed: Had to Swallow Med More Than Once | 2
  Agreed: Had to Swallow Med More Than Once | 5

4. Primary Outcome: Number of Participants Who Successfully Swallowed Study Med on Day 9
Description: The Swallowing Ability Questionnaire was completed on Day 9 after the participant received two matching placebo tablets (excluding marking) following consumption of a low- to moderate-fat meal in pediatric participants aged 10 to 17 years. The questionnaire consisted of five parts: could only swallow study med with help, easy to start swallowing study med, easy to swallow study med, felt like study med got stuck in throat, and had to swallow study med more than once. The number of participants who strongly agreed or agreed in each of the five parts is reported.
Time Frame: Day 9
Population: Per protocol population defined as all participants who completed at least one period of treatment and had available data. On Day 9, all participants received matching placebo, so the two treatment groups were pooled on Day 9.
Measure: Number; unit: Participants
Groups:
- All Treated Participants: All participants who completed at least one period of treatment and had available data. All participants received a single dose of two matching placebo tablets on Day 9.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 24
Participants
  Strongly Agreed: Could Only Swallow Med With Help | 9
  Agreed: Could Only Swallow Med With Help | 5
  Strongly Agreed: Easy to Start Swallowing Med | 9
  Agreed: Easy to Start Swallowing Med | 13
  Strongly Agreed: Easy to Swallow Med | 12
  Agreed: Easy to Swallow Med | 11
  Strongly Agreed: Felt Like Med Got Stuck in Throat | 1
  Agreed: Felt Like Med Got Stuck in Throat | 1
  Strongly Agreed: Had to Swallow Med More Than Once | 2
  Agreed: Had to Swallow Med More Than Once | 5

5. Primary Outcome: Area Under the Curve 0 to Last (AUC 0-last) of Sitagliptin Following Single Administration of Sitagliptin/Metformin XR
Description: In this study, metformin products were withheld 24 hours (hrs) prior to sitagliptin/metformin XR administration and were permitted to re-initiate 24 hrs post study drug administration. Owing to resumption of therapeutic metformin administration 24 hrs after sitagliptin/metformin XR administration for all participants, metformin pharmacokinetic analyses were restricted to maximum plasma concentration (Cmax), time to maximum plasma concentration (Tmax) and area under the curve 0 to 24 hrs (AUC0-24hr). Therefore, metformin arm is not included in this endpoint.
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, and 72 hours post-dose
Population: Per protocol population defined as all participants who completed at least one period of treatment (Sitagliptin/Metformin XR Followed by Placebo arm) and had available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr/mL
Groups:
- Sitagliptin: Day 1 (Period 1): participants received a single dose of two sitagliptin/metformin XR tablets with a low- to moderate-fat meal (breakfast). Days 2-4 (Period 1): participants received a single dose of two matching placebo tablets. Days 5-9 (Period 2): participants received a single dose of two matching placebo tablets with the evening meal.
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
nM*hr/mL | 5940 (25.7)

6. Primary Outcome: AUC 0-24 of Sitagliptin Following Single Administration of Sitagliptin/Metformin XR
Description: Due different units of measure for sitagliptin and metformin, metformin data are presented in another endpoint.
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, and 24 hours post-dose
Population: Per protocol population defined as all participants who completed at least one period of treatment and had available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
nM*hr | 5310 (22.4)

7. Primary Outcome: AUC 0-24 of Metformin Following Single Administration of Sitagliptin/Metformin XR
Description: In this study, metformin products were withheld 24 hours prior to sitagliptin/metformin XR administration and were permitted to re-initiate 24 hours post study drug administration. Due different units of measure for sitagliptin and metformin, sitagliptin data are presented in another endpoint.
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, and 24 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Metformin: Day 1 (Period 1): participants received a single dose of two sitagliptin/metformin XR tablets with a low- to moderate-fat meal (breakfast). Days 2-4 (Period 1): participants received a single dose of two matching placebo tablets. Days 5-9 (Period 2): participants received a single dose of two matching placebo tablets with the evening meal.
Arm/Group | Metformin
Number analyzed (Participants) | 12
ng*hr/mL | 14200 (39.7)

8. Primary Outcome: Area Under the Curve 0 to Infinity (AUC 0-∞) of Sitagliptin Following Single Administration of Sitagliptin/Metformin XR
Description: In this study, metformin products were withheld 24 hours prior to sitagliptin/metformin XR administration and were permitted to re-initiate 24 hours post study drug administration. Owing to resumption of therapeutic metformin administration 24 hours after sitagliptin/metformin XR administration for all participants, metformin pharmacokinetic analyses were restricted to Cmax, Tmax and AUC0-24hr. Therefore, metformin arm is not included in this endpoint.
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
nM*hr | 6020 (24.8)

9. Primary Outcome: Cmax of Sitagliptin Following Single Dose Administration of Sitagliptin/Metformin XR
Description: Due different units of measure for sitagliptin and metformin, metformin data are presented in another endpoint.
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
nM | 757 (40.1)

10. Primary Outcome: Cmax of Metformin Following Single Dose Administration of Sitagliptin/Metformin XR
Description: as for outcome 7
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Metformin
Number analyzed (Participants) | 12
ng/mL | 1490 (29.1)

11. Primary Outcome: Tmax of Sitagliptin and Metformin Following Single Dose Administration of Sitagliptin/Metformin XR
Description: In this study, metformin products were withheld 24 hours prior to sitagliptin/metformin XR administration and were permitted to re-initiate 24 hours post study drug administration.
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: Hour
Arm/Group | Sitagliptin | Metformin
Number analyzed (Participants) | 12 | 12
Hour | 1.52 [0.97 to 3.05] | 5.00 [3.98 to 7.22]

12. Primary Outcome: Apparent Terminal Half Life (t1/2) of Sitagliptin Following Single Dose Administration of Sitagliptin/Metformin XR
Description: as for outcome 8
Time Frame: Pre-dose, and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
Hour | 10.0 (27.3)

13. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Up to 23 days (including approximately 10 to 14 days after the last dose of study drug)
Population: All participants as treated defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 5 | 5

14. Primary Outcome: Number of Participants Who Experienced an Abnormal Vital Sign Value
Description: Vital sign measurements included blood pressure, heart rate, respiratory rate, and oral temperature.
Time Frame: Up to 23 days (including approximately 10 to 14 days after the last dose of study drug)
Population: All participants as treated defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

15. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Time Frame: Up to 9 days
Population: All participants as treated defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 23 days (including approximately 10 to 14 days after the last dose of study drug)
Description: All participants as treated defined as all participants who received at least one dose of study drug.
Arm/Group | Sitagliptin/Metformin XR Followed by Placebo | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Metformin XR Followed by Placebo (N=13) | Placebo (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.